CLINICAL TRIAL: NCT05382117
Title: Cardiac Rhythm and Affecting Factors in Patients Hospitalized in the Physical Therapy and Rehabilitation Clinic
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Hande Ozdemir, Assoc. Prof., Trakya University
Other Study IDs: 2021/161
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Neurumusculoskeletal Disorders
Keywords: neuromusculoskeletal, cardiovascular fitness,rhythm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In our study, it is aimed to evaluate the cardiac rhythms of patients who are decided to receive inpatient treatment in the physical therapy and rehabilitation clinic due to any neuromusculoskeletal diseases with 24 hour rhythm holter follow up on the day of hospitalization and three weeks after hospitalization and to determine the factors that may affect this result if a significant change is observed between the two measurements.The present results will guide the determination of the exercise duration, intensity, type and severity of the exercises to be created within the scope of the treatment programs of the patients and will lead to similar studies.

DETAILED DESCRIPTION:
Neuromusculoskeletal disorders include a variety of fairly common pathologies that can have a major impact on a person's health. Today, neuromusculoskeletal diseases are the main causes of occupational diseases and chronic physical disability leading to high health care costs globally. Exercise therapy is seen as an important part of the treatment of many neuromusculoskeletal diseases.

Patients hospitalized in the physical therapy and rehabilitation clinic are generally elderly people with chronic neuromusculoskeletal system disorders. While the presence of ventricular premature beat is detected in more than 50% of healthy adults in 24 hour rhythm holter examination, this rate rises above 90% in the elderly.Although many studies have noted that regular exercise and high cardiovascular fitness reduce the risk of cardiovascular arrhythmias, exercise may paradoxically increase the risk of sudden cardiac death in those with preexisting cardiac abnormalities.

There are no studies evaluating the changes in heart rhythms during hospitalization of patients hospitalized for treatment in physical therapy and rehabilitation clinics where exercise therapy is frequently applied.In our study, it is aimed to evaluate the cardiac rhythms of patients who receive inpatient treatment in the physical therapy and rehabilitation clinic with 24 hour rhythm holter follow up on the day of hospitalization and three weeks after hospitalization and to determine the factors that may affect this result if a significant change is observed between the two measurements.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old
* To be evaluated for any neuromusculoskeletal system disease and decided to be treated as an inpatient in the physical therapy and rehabilitation clinic
* Having agreed to participate in the study

Exclusion Criteria:

* A change in medication that may affect cardiac rhythm in the last two weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in Trakya University Hospital Physiotherapy and Rehabilitation Clinic
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-12-29 (Actual); Primary Completion 2022-12-28 (Estimated); Study Completion 2022-12-28 (Estimated)

PRIMARY OUTCOMES:
Evalution of the cardiac arrhythmia | up to three weeks
  24-hour cardiac rhythm recording by holter device

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University Medical Faculty, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robinson JG, Bakris G, Torner J, Stone NJ, Wallace R. Is it time for a cardiovascular primary prevention trial in the elderly? Stroke. 2007 Feb;38(2):441-50. doi: 10.1161/01.STR.0000254602.58896.d2. Epub 2006 Dec 28. PMID 17194877
- [Background] Ephrem G, Levine M, Friedmann P, Schweitzer P. The prognostic significance of frequency and morphology of premature ventricular complexes during ambulatory holter monitoring. Ann Noninvasive Electrocardiol. 2013 Mar;18(2):118-25. doi: 10.1111/anec.12010. Epub 2012 Nov 22. PMID 23530481
- [Background] Winkens RA, Hoppener PF, Kragten JA, Verburg MP, Crebolder HF. Are premature ventricular contractions always harmless? Eur J Gen Pract. 2014 Jun;20(2):134-8. doi: 10.3109/13814788.2013.859243. Epub 2013 Nov 28. PMID 24286118
- [Background] Frishman WH, Heiman M, Karpenos A, Ooi WL, Mitzner A, Goldkorn R, Greenberg S. Twenty-four-hour ambulatory electrocardiography in elderly subjects: prevalence of various arrhythmias and prognostic implications (report from the Bronx Longitudinal Aging Study). Am Heart J. 1996 Aug;132(2 Pt 1):297-302. doi: 10.1016/s0002-8703(96)90425-1. PMID 8701890
- [Background] Morris JN, Heady JA, Raffle PA, Roberts CG, Parks JW. Coronary heart-disease and physical activity of work. Lancet. 1953 Nov 28;262(6796):1111-20; concl. doi: 10.1016/s0140-6736(53)91495-0. No abstract available. PMID 13110075
- [Background] Harmon KG, Drezner JA, Wilson MG, Sharma S. Incidence of sudden cardiac death in athletes: a state-of-the-art review. Heart. 2014 Aug;100(16):1227-34. doi: 10.1136/heartjnl-2014-093872.rep. PMID 25049314
- [Background] Adrian D. Elliott , Dominik Linz, Christian V. Verdicchio, Prashanthan Sanders Centre for Heart Rhythm Disorders, University of Adelaide, Royal Adelaide Hospital and the South Australian Health & Medical Research Institute, 7 Adelaide, SA, Australia Heart, Lung and Circulation (2018) xx, 1--8 1443-9506/04
- [Background] Lewczuk J, Piszko P, Jagas J, Porada A, Sobkowicz-Wozniak B, Wrabec K. [Effect of acute exercise on cardiac arrhythmias in the course of chronic obstructive pulmonary disease]. Pneumonol Alergol Pol. 1994;62(9-10):496-500. Polish. PMID 7866322
- [Background] Manolis AS, Manolis AA. Exercise and Arrhythmias: A Double-Edged Sword. Pacing Clin Electrophysiol. 2016 Jul;39(7):748-62. doi: 10.1111/pace.12879. Epub 2016 May 25. PMID 27120033